CLINICAL TRIAL: NCT03792074
Title: to Evaluate SCT510 Compared to Avasitin Respectively Combined Paclitaxel and Carboplatin First-line Treatment of Locally Advanced and Metastatic or Recurrent Squamous Cell Non-small Cell Lung Cancer Efficacy and Safety
Brief Title: To Evaluate the Efficacy and Safety of SCT510 in the Treatment of Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCT510-A301
Record Dates: First submitted 2018-12-26; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Non-squamous Cell Non-small Cell Lung Cancer
MeSH Terms: interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCT510 combined paclitaxel and carboplatin (Experimental): SCT510 15mg/kg+ paclitaxel 175mg+ carboplatin (AUC=5), intravenous infusion，on day 1，Once every 3 weeks;Four to six cycles in a row
  Interventions: Drug: SCT510; Drug: Paclitaxel; Drug: Carboplatin
- Bevacizumab combined paclitaxel and carboplatin (Active Comparator): Bevacizumab 15mg/kg+ paclitaxel 175mg+ carboplatin (AUC=5), intravenous infusion，on day 1，Once every 3 weeks;Four to six cycles in a row
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: SCT510 — SCT510 Injection
  Arms: SCT510 combined paclitaxel and carboplatin
Drug: Bevacizumab — Bevacizumab Injection
  Other Names: Avastin
  Arms: Bevacizumab combined paclitaxel and carboplatin
Drug: Paclitaxel — Paclitaxel Injection
  Other Names: PTX;TAX
Drug: Carboplatin — Carboplatin injection

SUMMARY:
To evaluate the safety, efficacy and immunogenicity of SCT510 combined with paclitaxel and carboplatin compared with bevacizumab combined with paclitaxel and carboplatin in the first-line treatment of locally advanced metastatic or recurrent squamous cell non-small cell lung cancer.

DETAILED DESCRIPTION:
A randomized, double-blind, parallel-controlled, multicenter phase 3 clinical trial.

560 patients with non-resectable locally advanced, metastatic or recurrent non-squamous cell non-small cell lung cancer (NSCLC) were randomly divided into two groups (SCT510 group and bevacizumab group) at a 1:1 ratio, and the treatment included combination chemotherapy and maintenance treatment, followed by follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this study and sign the informed consent;
2. age is ≤ 18 years old and ≥ 80 years old, regardless of gender;
3. Subjects with unresectable locally advanced metastatic（Not suitable for the multidisciplinary treatment Ⅲ B - Ⅳ period of subjects, according to the international association for the study of lung cancer (IASLC) lung cancer staging manual version 8 standard judgment） or recurrent non-squamous cell non-small cell lung cancer diagnosed by histological and/or cytological examination.The diagnosis of non-squamous cell non-small cell lung cancer based on sputum cytology requires immunohistochemical confirmation.If multiple tumor components are mixed, the main cell types are classified.
4. It is able to provide relevant documents about EGFR mutation and ALK fusion gene status, and there is no EGFR sensitive mutation (including exon mutation no. 18 (G719X), exon deletion no. 19 and exon mutation no. 21 (L858R, L861Q)) and ALK fusion.Subjects who have not previously undergone EGFR and ALK gene testing will need to undergo genetic testing during the screening period.Among them, subjects whose EGFR or ALK gene status cannot be determined for various reasons can be enrolled;Subjects who are known to have EGFR sensitive mutations and/or ALK fusion may also be enrolled if they are currently unable to obtain the corresponding targeted drugs (including the rejection of the subjects) and chemotherapy is standard treatment at the research center;
5. According to RECIST v1.1 criteria, at least one measurable lesion was ensured;The lesions that had received radiotherapy before could only be selected as target lesions if there was clear disease progression 3 months after the end of radiotherapy.
6. Systemic antitumor therapy for locally advanced metastatic or recurrent non-squamous non-small cell lung cancer has not been accepted.If the subjects in the complete early non-small cell lung cancer after radical treatment received adjuvant therapy, and disease relapse, participants need to ensure that adjuvant therapy over time from this study first dosing interval more than 6 months, and auxiliary treatment led to a variety of toxic effects have been restored (according to the CTCAE v4.03 standard judgment level 1 or less, except for hair loss).
7. Eastern Cooperative Oncology Group （ECOG） physical condition score 0 or 1
8. the expected survival time is more than 6 months;
9. Laboratory inspection meets the following requirements:

   * absolute neutrophil value (ANC) is greater than 1.5 x 109/L, platelet count (PLT) is greater than 100 x 109/L, hemoglobin (HGB) is greater than 90 g/L, and white blood cell (WBC) is greater than 3.0 x 109/L;
   * liver function: total bilirubin (TBil) < 1.5 times the normal upper limit; Aspartate aminotransferase(AST/SGOT),Alanine aminotransferase (ALT/SGPT),andalkaline phosphatase(ALP) < 2.5 times the normal upper limit;In the case of liver metastasis, AST and ALT were less than or equal to 5.0 times the upper limit of normal values.In the case of liver metastasis and/or bone metastasis, ALP is less than or equal to 5.0 times the normal upper limit.
   * renal function: upper limit of normal serum creatinine (Scr) less than 1.5 times;
   * urine protein < 2 (+) detected by routine urine test;If the urine protein at baseline is greater than or equal to 2 (+), the 24-hour urine protein quantification must be less than or equal to 1.0 g.
   * coagulation function: the international standardized ratio (INR) is no more than 1.5, and the activation time of partial thrombin (APTT) is no more than 1.5 times the upper limit of normal value;
10. Heart function: left ventricular ejection fraction (LVEF) 50% or higher;
11. able to communicate well with researchers and follow the visit, treatment, laboratory examination and other relevant regulations stipulated in the study.

Exclusion Criteria:

1. subjects with mixed non-small cell and small cell carcinoma, squamous cell carcinoma or mixed adenosquamous carcinoma with squamous cell as the main component
2. patients with a history of tracheoesophageal fistula, gastrointestinal perforation or gastrointestinal fistula and intraperitoneal abscess within 6 months before randomization;
3. patients with malignant tumors other than lung cancer within the first 5 years were randomized, excluding cured carcinoma in situ of the cervix, skin basal cells cancer or squamous epithelial cells skin cancer, local prostate cancer after radical resection and ductal carcinoma in situ of the breast after radical resection;
4. severe cardiovascular and cerebrovascular diseases, including cerebrovascular accidents (CVA), transient ischemic attack (TIA), myocardial infarction and significant vascular diseases (including but not limited to aortic aneurysms requiring surgical repair or recent arterial thrombosis) within the first 6 months randomly;Patients with unstable angina, New York heart association (NYHA) classification ≥ Ⅱ heart failure and arrhythmia drugs can't control;
5. Subjects who received lung radiotherapy within the first 4 weeks or who had not recovered from radiation-related toxicity were randomized.For all other anatomical sites, subjects received radiotherapy within the first 2 weeks of randomization or did not recover from radiation-related toxicity;
6. Major surgery was performed within the first 4 weeks of randomization or major surgical treatment was planned during the trial period (the researchers determined that there was a risk of bleeding or wound healing complications);
7. Have bleeding tendency, high bleeding risk or coagulation dysfunction, including thrombotic disease within 6 months prior to randomization and/or hemoptysis history within 3 months prior to randomization (single hemoptysis is more than 2.5mL);Or recently (less than 10 days after the first study drug treatment) using a full dose oral or extralimental anticoagulant or thrombolytic agent or aspirin (> 325 mg/ day) or other nsaids that inhibit platelet function;Or prior to surgery, the researchers determined that there was a tendency to bleed;
8. subjects with high suspicion of idiopathic pulmonary fibrosis, organic pneumonia, drug-related pneumonia, idiopathic pneumonia or active pneumonia in chest CT scan during the screening period;
9. subjects with known central nervous system metastasis (except asymptomatic brain metastasis and subjects with treated symptoms controlled and stable symptoms within 1 month prior to randomization).Patients with clinical suspected central nervous system metastasis must undergo enhanced CT or MRI within the first 28 days randomly to exclude central nervous system metastasis.
10. imaging examination showed signs of tumor invasion into the large blood vessel, and the tumor had completely approached, wrapped or invaded the large blood vessel cavity (such as pulmonary artery or superior vena cava);
11. patients with hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg) who are still under poor control after combined treatment with two or more antihypertensive drugs in the screening period, as well as those who have a history of hypertension crisis or hypertensive encephalosis;
12. The presence of unhealed wounds, active peptic ulcers and fractures (excluding healed old fractures);
13. There is a large amount of pericardial effusion, peritoneal or pleural effusion that cannot be controlled by drainage or other symptomatic treatment (symptomatic treatment is allowed before enrollment, but drugs with anti-tumor indications, such as chemotherapy drugs, anti-angiogenic drugs and molecular targeted drugs, cannot be given);
14. HBsAg is positive, and the titer detection of HBV-DNA in peripheral blood ≥ 1x103 copy number /mL (or the quantitative determination of HBV-DNA ≥200 units /mL); HCV or HIV or syphilis positive subjects;At present, there are other active infectious diseases, which are not suitable for inclusion in this study.
15. known for SCT510, bevacizumab, paclitaxel and carboplatin injection and its material composition allergies;
16. women who are pregnant or breast-feeding;
17. women of child-bearing age or male subjects who are unwilling to take effective contraceptive measures during the study period or within 6 months after the last administration of the study drugs;
18. subjects who have participated in other clinical studies in the first 4 weeks of randomization or who are receiving treatment in other clinical trials (except those who participated in the overall survival follow-up of one study);
19. previous history of alcoholism or drug abuse;
20. in addition to the above circumstances, the researcher believes that there are other circumstances that are not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 12 weeks
  the proportion of subjects whose CR（complete response） and PR（partial response）combined , according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Objective response rate | 18 week
  the proportion of subjects whose CR（complete response） and PR（partial response）combined , according to RECIST 1.1 criteria
Disease control rate | 12 weeks and 18 weeks
  the proportion of subjects with CR（complete response）, PR（partial response） and SD（Stable disease） combined，according to RECIST 1.1 criteria
Duration of Response | 3 years
  The time from the first assessment of CR（complete response） or PR（partial response） to the first assessment of PD（progressive disease） or any cause of death，according to RECIST 1.1 criteria
Progression free survival | 3 years
  The time from randomization to PD（progressive disease） or any cause of death，according to RECIST 1.1 criteria
1-year overall survival rate | 1 year
  The proportion of subjects who survived longer than 1 year after randomization
Overall survival | 3 years
  Defined as the time from randomization of subjects to death from any cause

REFERENCES:
- [Derived] Hong Q, Jiao Y, Li D, Ma H, Wu K, Xie L. Population Pharmacokinetics of SCT510 (a Bevacizumab Biosimilar) and Avastin(R) in Healthy Subjects and Patients with Non-squamous Non-small Cell Lung Cancer. Clin Drug Investig. 2026 Feb;46(2):143-157. doi: 10.1007/s40261-025-01518-8. Epub 2026 Jan 6. PMID 41495391
- [Derived] Cheng Y, Pan Z, Wu L, Zhu B, Yu Y, Zang K, Zhuang W, Liu L, Gu K, Lian J, Chen R, Bian T, Lin D, Sun S, Li W, Hang X, Jiang O, Zhong F, Wang R, Luo H, Shi H, Wei Z, Zhao L, Chen S, Sun H, Li X, Sun D, Ren T, Lei K, He M, Li G, Liu H, Li R, Hu C, Kong L, Sun M, Xie L, Gai W, Chen W, Huang Z, Ren W, Su H. Efficacy and Safety of Biosimilar SCT510 Compared with Bevacizumab for the First-Line Treatment of Advanced Non-Squamous Non-Small Cell Lung Cancer: A Randomized, Double-Blind, Phase III Study. Adv Ther. 2024 Nov;41(11):4032-4048. doi: 10.1007/s12325-024-02965-z. Epub 2024 Sep 4. PMID 39230871